CLINICAL TRIAL: NCT04491214
Title: Post ICU Follow up in Patients With Severe SARS-CoV-2 Infection (Covid-19)
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7890
Record Dates: First submitted 2020-07-20; First posted 2020-07-29 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2020-02

CONDITIONS: Covid19; Follow up; Rehabilitation
Keywords: SARS-CoV-2; Follow up; Intensive care unit; Cohort
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: quality of live assessment — quality of live assessment 3 moth and 6 moth after ointensive care hospitalisation using SF36.

SUMMARY:
Patients affected by new coronavirus infectious disease (COVID) were mostly hospitalized in ICU. This infection seems to cause widespread organ injury (i.e acute renal injury, neurological disorders, pulmonary embolism,…). It is therefore necessary to provide a framework for the follow up of patients. Moreover SARS-CoV-2 infection consequences remain unknow at this time. Study hypothesis is that COVID alters determining factors (physical or psychological) of quality of life after ICU hospitalisation. The aim of the study is to assess quality of life 3 months after ICU hospitalization.

Secondary purposes of the study are 1) assessment of quality of life 6 months and the evolution between the third and the sixth months after ICU hospitalization 2) description patients care after 3 and 6 months ICU left and their clinical status 3) convening and providing a "platform" within several physicians (neurologist, biologist, pneumologist…) will be able to follow up patients and perform complementary investigations according to patients injuries.

ELIGIBILITY:
Inclusion criteria:

* Subject male or female ≥ 18 years old
* Patient hospitalized in the anesthesia-resuscitation department of the NHC for COVID-19 from March 1, 2020.
* Patient (or his legal representative) having given his consent for the use of his data for the purposes of this research.

exclusion criteria:

* Subject not hospitalized in intensive care
* Patient's refusal to participate in the study
* Inability to give informed information to the subject (subject in an emergency, difficulty understanding the subject, etc.)
* Subject under low protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with severe SARS-Cov-2 hospitalized in intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
assess quality of life after severe COVID infection | measured at 3 months after ICU left.
  assess different dimensions of quality of life: physical and mentaland social dimensions

SECONDARY OUTCOMES:
Quality of life and Clinical status | measured at 3 and 6 months after ICU left.
  Clinical status of patients and assessment of quality of life. collects crucial elements of care based on doctors' prescriptions

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg (Nouvel Hôpital Civil), Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided